CLINICAL TRIAL: NCT07065487
Title: Accuracy of Standard vs Geometric Pattern-Assisted Digital Scanning Techniques for Construction of Full Arch Implant Prosthesis Framework: A Crossover Study
Brief Title: Accuracy of Standard and Geometric Pattern-Assisted Digital Scanning for Full-Arch Implant Prosthesis Frameworks
Acronym: GPA Scan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mirna ashraf anis heneen (Other)
Responsible Party: Sponsor-Investigator, Mirna ashraf anis heneen, Assistant Lecturer of Prosthodontics, Horus University, Damietta - PhD Candidate, Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MU-PROS-2025-001
Record Dates: First submitted 2025-06-20; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Edentulous Jaw; Dental Prosthesis, Implant-Supported; Prosthodontics; Dental Implantation, Endosseous
Keywords: Digital impression; Full-arch implant; Geometric pattern; Prosthesis framework; Intraoral scanner; Splinted impression; CAD/CAM prosthodontics; Passive fit; Dental implants
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: randomized crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Splinted Impression (Experimental): Participants will undergo a conventional impression technique using open-tray impression copings rigidly splinted with DuraLay resin. The impression is taken using polyvinyl siloxane (PVS) material in a custom tray. This method serves as the control for comparison with digital techniques.
  Interventions: Procedure: Conventional Splinted Impression Technique
- Standard Digital Scan (Experimental): Participants will undergo a full-arch digital scan using an intraoral scanner. Scan bodies will be attached to the multi-unit abutments, and the scan will be performed without any additional geometric reference aids.
  Interventions: Device: Intraoral Scanner - Standard Protocol
- Geometric Pattern-Assisted Digital Scan (Experimental): Participants will undergo a full-arch digital scan using an intraoral scanner, with the addition of a geometric reference pattern placed in the scanning field to improve stitching accuracy and scan reliability.
  Interventions: Device: Intraoral Scanner with Geometric Reference Pattern

INTERVENTIONS:
Device: Intraoral Scanner - Standard Protocol — A full-arch digital impression is obtained using a high-precision intraoral scanner. Scan bodies are placed on multi-unit abutments and scanned without the use of external reference markers or geometric aids. The scan follows the manufacturer-recommended scanning path to capture the complete arch. This serves as a baseline digital technique for comparison with geometric pattern-assisted scanning.
  Arms: Standard Digital Scan
Device: Intraoral Scanner with Geometric Reference Pattern — The same intraoral scanner is used, but with an additional geometric reference pattern introduced in the scanning field to improve stitching accuracy and alignment of the digital scan.
  Arms: Geometric Pattern-Assisted Digital Scan
Procedure: Conventional Splinted Impression Technique — A physical impression is taken using open-tray impression copings splinted with DuraLay resin and polyvinyl siloxane (PVS) material in a custom tray, according to conventional protocols for full-arch implant prostheses.
  Arms: Conventional Splinted Impression

SUMMARY:
This clinical trial aims to compare three different impression techniques used to fabricate full-arch implant-supported dental prostheses. Accurate impressions are essential to ensure a passive and precise fit of the final prosthetic framework, which contributes to long-term implant success and patient comfort.

In this crossover study, participants with four osseointegrated dental implants in the lower jaw will undergo three types of impressions:

Conventional splinted impression using polyvinyl siloxane (PVS) material.

Standard digital impression using an intraoral scanner.

Geometric pattern-assisted digital impression, which incorporates a visual reference pattern to improve scan alignment and accuracy.

Each participant will receive all three impression techniques in a randomized sequence, at different time points. The accuracy of each method will be assessed by evaluating the passivity of the resulting prosthetic frameworks using two methods: (1) digital superimposition analysis to measure three-dimensional (3D) spatial deviation, and (2) the clinical "one-screw test" to detect misfit.

The study seeks to determine whether digital scanning, particularly with geometric pattern assistance, can provide accuracy comparable to or better than conventional methods. Findings may guide improvements in digital prosthodontic workflows and support more efficient, predictable treatment outcomes.

DETAILED DESCRIPTION:
This is a prospective, crossover clinical trial designed to evaluate and compare the accuracy of three different impression techniques used in the fabrication of full-arch implant-supported prosthesis frameworks. The study includes four participants, each with four osseointegrated dental implants in the mandibular arch.

The three impression techniques being compared are:

Conventional Splinted Impressions: A traditional method utilizing rigidly splinted impression copings and polyvinyl siloxane (PVS) impression material to capture implant positions.

Standard Digital Scanning: A fully digital technique using an intraoral scanner and scan bodies placed on the implants to generate a digital impression.

Geometric Pattern-Assisted Digital Scanning: An enhanced digital method incorporating a geometric reference pattern during the scanning process to improve stitching accuracy and reduce scan distortion across the arch.

Each participant will receive all three impression techniques in a randomized sequence to minimize order bias. Digital models will be generated from each impression method, and test frameworks will be designed using computer-aided design/computer-aided manufacturing (CAD/CAM) technology. These frameworks will be fabricated using 3D laser sintering.

The primary outcome of the study is the assessment of accuracy, defined as the mean three-dimensional (3D) deviation between the test scan and a reference scan, measured via digital superimposition software. A secondary outcome is clinical passivity, evaluated using the one-screw test to detect any misfit between the framework and implant interfaces.

The results of this study aim to provide clinical evidence regarding the accuracy and feasibility of advanced digital impression techniques, particularly the use of geometric pattern references, in full-arch implant prosthodontics. This may support improvements in digital workflow reliability, patient outcomes, and prosthetic longevity.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 30 to 70 years

Completely edentulous mandible

Presence of four osseointegrated implants in the lower jaw

Good oral and general health

Willingness to participate and provide written informed consent

Availability for all study appointments

Exclusion Criteria:

Systemic diseases or conditions that affect bone healing or implant integration

Presence of oral inflammation, infection, or soft tissue abnormalities at implant sites

History of bruxism or parafunctional habits

Inability to understand or comply with study procedures

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Mean 3D deviation (in microns) between test and reference scans using digital superimposition. | Immediately after each impression session (Day 0 for each method).
  Accuracy will be assessed by digitally superimposing the scan obtained from each method (conventional splinted impression, standard digital scan, geometric pattern-assisted digital scan) onto a reference scan (conventional method). Specialized software will calculate the mean 3D deviation in microns to quantify spatial accuracy. Lower deviation indicates higher accuracy.

SECONDARY OUTCOMES:
Number of frameworks exhibiting passive fit as determined by the one-screw test. | Within 1 hour of framework placement following each impression method.
  Clinical assessment of framework passivity will be performed using the one-screw test. A passive fit will be recorded if no lifting or rocking is observed upon tightening a single screw at one end of the framework while the others remain untightened. Count and percentage of frameworks with passive fit will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including digital scan accuracy values and framework fit results, will be made available upon reasonable request after publication of the study results. Data will be shared with qualified researchers for academic and non-commercial purposes only, subject to ethical approval and data-sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after publication of the study results and for up to 5 years.
Access Criteria: De-identified individual participant data (IPD) and supporting materials (study protocol, statistical analysis plan, and informed consent form) will be available to qualified researchers affiliated with academic institutions or non-profit organizations. Access will be granted for non-commercial, ethically approved research purposes. Interested researchers must submit a formal request to the Principal Investigator via email, including a research proposal and institutional ethical approval. Access will be provided through secure, password-protected file sharing platforms.